CLINICAL TRIAL: NCT06982729
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of YK012 in the Treatment of Primary Membranous Nephropathy
Brief Title: Study of YK012 in Primary Membranous Nephropathy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Excyte Biopharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YK012-3-CN
Record Dates: First submitted 2025-05-06; First posted 2025-05-21 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Primary Membranous Nephropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ia: YK012 (Experimental): Participants with primary membranous nephropathy will receive ascending doses of YK012 infusion to evaluate the safety and tolerability of YK012
  Interventions: Drug: YK012
- Ib: YK012 (Experimental): Participants will receive 2 different doses of YK012 infusion to assess the preliminary efficacy of YK012 in participants with primary membranous nephropathy and to establish the recommended Phase II dose (RP2D).
  Interventions: Drug: YK012

INTERVENTIONS:
Drug: YK012 — YK012 is a bispecific antibody targeting CD19 on B cells and CD3 on T cells leading to T cell-mediated cytotoxicity of malignant B cells
  Other Names: YK012 Infusion

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), immunogenicity, and preliminary efficacy of YK012 in participants with primary membranous nephropathy (PMN).

DETAILED DESCRIPTION:
This clinical trial consists of Phase Ia and Phase Ib. The goal of phase Ia is to evaluate the safety and tolerability of YK012 in participants with primary membranous nephropathy and to determine the maximum tolerated dose (MTD) and recommended dose for expansion (RDE). The goal of phase Ib is to assess the preliminary efficacy of YK012 in participants with primary membranous nephropathy and to establish the recommended Phase II dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years (inclusive), regardless of gender.
* Kidney biopsy-confirmed diagnosis of primary (idiopathic) membranous nephropathy within the past 10 years.
* Elevated 24-hour urine protein, meeting the pre-defined criteria.
* Estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73m² as calculated by the CKD-EPI equation.
* If currently taking an angiotensin-converting enzyme inhibitor (ACEi), angiotensin II receptor blocker (ARB), or sodium-glucose cotransporter-2 (SGLT-2) inhibitor, the dose must have been stable for at least 4 weeks prior to enrollment or since initiation of therapy.
* Laboratory test results must meet the predefined criteria within 7 days prior to enrollment.
* Capable of understanding and voluntarily participating in this clinical trial, having provided written informed consent, and able to comply with scheduled visits, treatments, examinations, and other study procedures as required.

Exclusion Criteria:

* Diagnosis of secondary membranous nephropathy.
* Any prior receipt of protocol-specified pharmacological treatment for membranous nephropathy.
* History of malignancy within 5 years prior to enrollment.
* Poorly controlled hypertension at enrollment.
* Severe renal dysfunction with prior dialysis or kidney transplantation within 6 months prior to enrollment.
* Prior kidney biopsy-confirmed diagnosis of diabetic nephropathy.
* History of severe or chronic infections within the 6 months before enrollment or current need for systemic antibiotic or antiviral therapy.
* Cardiovascular or cerebrovascular events requiring hospitalization within 6 months prior to enrollment.
* Severe or poorly controlled comorbidities that may affect protocol compliance or efficacy evaluation.
* Active Tuberculosis (TB) with documented evidence of infection.
* History of solid organ or bone marrow transplantation.
* Live vaccination, major surgery, or participated in other clinical trials with investigational drug use within 28 days prior to enrollment.
* HBsAg-positive, or HBcAb-positive with detectable HBV DNA above the normal range; HCV antibody-positive; HIV seropositive; Treponema pallidum antibody-positive.
* CD4+ T lymphocyte count <200 cells/μL
* Known hypersensitivity to any component of YK012.
* Pregnancy, breastfeeding, or positive pregnancy test at screening; or plans to become pregnant during the trial or within 12 months after study completion, or unwillingness to use physical contraceptive methods during the study and for 12 months thereafter.
* Other conditions deemed by the investigator to make the subject unsuitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Ia: Dose-limiting Toxicity(DLT) | up to 28 days after the first dose
  Dose-limiting toxicities (DLTs) is defined as adverse events occurring within 28 days after the first dose and assessed by the investigator as related to the Investigational Medicinal Product (IMP).
Ia: Adverse Event (AE) | From the first induction to the end of the trial at 53 weeks
  An AE is defined as any untoward medical event that occurs after a participant receives the investigational drug, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the investigational drug.
Ia: Severe Adverse Event | From the first induction to the end of the trial at 53 weeks
  An SAE refers to any untoward medical occurrence after the participant receives the IMP that results in one or more of the following: death, life-threatening event, permanent or serious disability or loss of function, hospitalization or prolongation of hospitalization, congenital abnormalities or birth defects.
Ib: Proportion of participants achieving overall response | From enrollment to the end of the trial at 76 weeks (if applicable)

SECONDARY OUTCOMES:
Ia: Area Under the Curve (AUC) of a serum concentration versus time profile | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
Ia: Area Under the Curve of a serum concentration to infinite time (AUC0-infinity) | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
Ia: Maximum concentration (Cmax) of YK012 | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
Ia: Time to reach Cmax (Tmax) | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
Ia: Elimination half life (t1/2) | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
Ia: Total Apparent Clearance (CL) | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
Ia: Apparent volume of distribution(Vd) | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
Ia: Minimum Concentration (Cmin) of YK012 | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
Ia: The duration of peripheral blood B-cell depletion | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
Ia: The profile of peripheral blood NK cell changes | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
Ia: The profile of peripheral blood T-cell changes | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
Ia: The profile of cytokine changes | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
Ia: ADA (anti-drug antibody) and Nab (Neutralizing antibody) positivity rate | From 1 hour before the first infusion of YK012 to the end of trial at 53 weeks
24-hour urine protein change | From enrollment to the end of the trial at 53 or 77 (if applicable) weeks
eGFR (Glomerular Filtration Rate) change | From enrollment to the end of the trial at 53 or 77 (if applicable) weeks
Anti-PLA2R antibody titer change | From enrollment to the end of the trial at 53 or 77 (if applicable) weeks
Ia: Proportion of participants achieving overall response | From enrollment to the end of the trial at 53 weeks
Proportion of participants achieving CR or PR | From enrollment to the end of the trial at 53 or 77 (if applicable) weeks
Proportion of anti-PLA2R antibody-positive participants achieving immunological remission | From enrollment to the end of the trial at 53 or 77 (if applicable) weeks
Time to achieve complete renal remission | From enrollment to the end of the trial at 53 or 77 (if applicable) weeks
Time to achieve overall renal response | From enrollment to the end of the trial at 53 or 77 (if applicable) weeks
Duration of complete renal response | From enrollment to the end of the trial at 53 or 77 (if applicable) weeks
Duration of overall renal response | From enrollment to the end of the trial at 53 or 77 (if applicable) weeks
Proportion of participants with treatment failure | From enrollment to the end of the trial at 53 or 77 (if applicable) weeks
Proportion of participants with relapse | From enrollment to the end of the trial at 53 or 77 (if applicable) weeks
Ib: Adverse Event (AE) | From the first induction to the end of the trial at 53 or 77 (if applicable) weeks
  An AE is defined as any untoward medical event that occurs after a participant receives the investigational drug, which may be manifested as symptoms, signs, diseases, or laboratory abnormalities, but may not necessarily have a causal relationship with the investigational drug.
Ib: Severe Adverse Event | From the first induction to the end of the trial at 53 or 77 (if applicable) weeks
  An SAE refers to any untoward medical occurrence after the participant receives the IMP that results in one or more of the following: death, life-threatening event, permanent or serious disability or loss of function, need for hospitalization or prolongation of hospitalization, congenital abnormalities or birth defects.

CONTACTS AND LOCATIONS:
Overall Officials: Minghui Zhao, M.D., Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China